CLINICAL TRIAL: NCT01004172
Title: Phase II Trial of Carboplatin and Bevacizumab for Progressive Breast Cancer Brain Metastases
Brief Title: Carboplatin and Bevacizumab for Progressive Breast Cancer Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nancy Lin, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-224
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Breast Cancer; Breast Cancer; Progressive Breast Cancer
Keywords: carboplatin; bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Bevacizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carboplatin, bevacizumab, trastuzumab (if HER2+) (Experimental): Participants received treatment until disease progression in either CNS or non-CNS site. Cycle duration is 28 days.
  carboplatin: AUC=5 dose given intravenously on day 8 of cycle one and Day 1 of each subsequent cycle
  bevacizumab: 15 mg/kg dose given intravenously on day 1 of each cycle
  trastuzumab*: 6 mg/kg dose given intravenously on day 8 of each cycle for patients with HER2-positive breast cancer only
  *8mg/kg loading dose in cycle 1 for some participants
  HER-2: human epidermal growth factor receptor 2
  Interventions: Drug: carboplatin; Drug: bevacizumab; Drug: herceptin

INTERVENTIONS:
Drug: carboplatin
Drug: bevacizumab
  Other Names: Avastin
Drug: herceptin
  Other Names: trastuzumab

SUMMARY:
The purpose of this research study is to determine how well the combination of bevacizumab and carboplatin works in treating breast cancer that has spread to the brain. Bevacizumab is an antibody (a protein that attacks a foreign substance in the body) that is made in the laboratory. Bevacizumab works differently from the way chemotherapy drugs work. Usually chemotherapy drugs attack fast growing cancer cells in the body. Bevacizumab works to slow or stop the growth of cells in cancer tumors by decreasing the blood supply to the tumors. When the blood supply is decreased, the tumors don't get the oxygen and nutrients they need to grow. Carboplatin is in a class of drugs known as platinum-containing compounds and has been approved for use in the treatment of ovarian cancer. Information from other research studies suggests that the combination of bevacizumab with carboplatin may be effective in treating breast cancer.

DETAILED DESCRIPTION:
This study used a two-stage design to evaluate efficacy bevacizumab and carboplatin based on Central Nervous System (CNS) response. The null and alternative therapy response rates are 5% versus 20%. If 1 or more participants assessable in the stage one cohort (n=12 assessable participants) achieve CNS response then accrual proceeds to stage two (n=25 additional assessable participants). If at least 4 participants in the final set of 37 assessable participants achieve CNS response then this regimen would be deemed worthy of further study. The probability of stopping early is 0.54 if the true CNS response rate is 5% and 0.07 if the true CNS response rate is 20%. The probability of deeming the treatment worthy of further study is 0.10 and 0.90 if the true CNS response rate is 5% and 20%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with metastatic disease. patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis by physical exam or radiologic study
* Measurable disease. Patients must have measurable CNS disease, defined as at least one parenchymal brain lesion that can be accurately measured in at least one dimension with longest dimension >/= 10mm by local radiology review
* New or progressive CNS lesions, as assessed by the patient's treating physician
* No increase in corticosteroid dose in the week prior to the baseline brain MRI
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group Performance Score (ECOG PS) performance status 0-2
* Normal organ and marrow function as outlined in the protocol
* Left ventricular ejection fraction >/= 50%, as determined by radionuclide ventriculography (RVG) or echocardiogram within 60 days prior to initiation of protocol therapy
* Prior carboplatin is allowed if it was not given in conjunction with bevacizumab
* Prior trastuzumab is allowed
* No prior bevacizumab since diagnosis of CNS metastases or within 6 months prior to diagnosis of CNS metastases
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Patients who have had chemotherapy within 14 days prior to entering the study, or those who have not recovered adequately from adverse events due to agents administered earlier
* Patients may not receive any concurrent investigational agents while on study
* Patients may not receive any cancer-directed concurrent therapy , such as concurrent chemotherapy, radiotherapy, or hormonal therapy while on study. Concurrent treatment with bisphosphonates is allowed
* History of Grade 3 or 4 allergic reactions attributed to compounds of similar or identical biologic composition to bevacizumab, carboplatin, or trastuzumab
* Known contraindication to MRI with gadolinium contrast, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Leptomeningeal carcinomatosis as the only site of CNS involvement
* More than 2 seizures over last 4 weeks prior to study entry
* Grade 1 or higher CNS hemorrhage on baseline brain MRI
* History of grade 2 or higher CNS hemorrhage within 12 months of study entry
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infraction or unstable angina within 6 months prior to day 1
* Significant vascular disease within 6 months prior to day 1
* History of hemoptysis within 1 month prior to day 1
* Evidence of bleeding diathesis or significant coagulopathy
* Current, ongoing treatment with full-dose warfarin or its equivalent
* Use of aspirin (>325 mg/day) within 10 days prior to day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 or anticipation of need for major surgical procedure during the course of the study.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a urine protein-creatinine ratio >/= 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leone JP, Emblem KE, Weitz M, Gelman RS, Schneider BP, Freedman RA, Younger J, Pinho MC, Sorensen AG, Gerstner ER, Harris G, Krop IE, Morganstern D, Sohl J, Hu J, Kasparian E, Winer EP, Lin NU. Phase II trial of carboplatin and bevacizumab in patients with breast cancer brain metastases. Breast Cancer Res. 2020 Nov 30;22(1):131. doi: 10.1186/s13058-020-01372-w. PMID 33256829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between November 2009 and August 2012.
Period: Overall Study
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Started | 38
Completed | 0
Not Completed | 38
Not completed — Progressive Disease in CNS Only | 16
Not completed — Progressive Disease in Non-CNS Only | 16
Not completed — Progressive Disease in CNS and Non-CNS | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Symptomatic Deterioration | 2

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
Age, Customized [Median (Full Range); unit: years] | 48 [31 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34
  Black or African-American | 1
  Asian | 3
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Objective Response Rate
Description: CNS objective response rate is the percentage of participants that achieve CNS complete or partial response as follows:
  CNS complete response (CR) is achieved if all of the following are satisfied:
  * Complete resolution of all measurable (>= 1 cm in longest dimension [LD]) and non-measurable brain metastases
  * No new CNS lesions (defined as any new lesion >= 6 mm in LD)
  * Stable or decreasing steroid dose
  * No new/progressive tumor-related neurologic signs or symptoms
  * No progression of extra-CNS disease as assessed by RECIST
  CNS partial response (PR) is achieved if all of the following are satisfied:
  ->/= 50% reduction in the volumetric sum of all measurable (>/= 1 cm in LD) brain metastases compared to baseline
  * No progression on non-measurable lesions
  * No new CNS lesions (defined as any new lesion >/= 6 mm in LD)
  * Stable or decreasing steroid dose
  * No new/progressive tumor-related neurologic signs or symptoms
  * No progression of extra-CNS disease as assessed by RECIST
Time Frame: Response was evaluated radiologically at baseline and every 2 cycles on treatment. Treatment duration for this study cohort was a median (range) of 8 cycles (1-20) which approximates months given the 4 week cycle length.
Population: The analysis dataset is comprised of assessable participants. Per protocol, assessable is defined as those who have at least one lesion on baseline MRI with longest with longest diameter >10 mm on T1-weighted, gadolinium-enhanced. All enrolled participants were assessable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
percentage of participants | 63 [47 to 77]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of disease progression (PD), second cancer, or death, whichever occurs first. PD if any of the following occur:
  CNS Disease
  * >/=40% increase in the volumetric sum of all measurable lesions as compared to the smallest volume on treatment
  * Progression of non-measurable lesions
  * New lesions (>/=6 mm)
  Non-CNS Disease
  • RECIST 1.0 criteria: at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded on treatment or the appearance of >/=1 new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
  Symptomatic
  * Increasing steroid requirement
  * Global deterioration of health status requiring discontinuation of treatment
  * New/progression tumor-related neurologic signs and symptoms except for transient worsening lasting </=14 days
Time Frame: Disease was evaluated radiologically at baseline, cycle 2, cycle 4 and thereafter on treatment every 2 cycles (CNS disease) and every 4 cycles (non-disease). Maximum PFS follow-up for this study cohort was 18.6 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carboplatin, Bevacizumab, Trastuzumab (if HER2+): Participants received treatment until disease progression in either CNS or non-CNS site. Cycle duration is 28 days.
  carboplatin: AUC=5 dose given intravenously on day 8 of cycle one and Day 1 of each subsequent cycle
  bevacizumab: 15 mg/kg dose given intravenously on day 1 of each cycle
  trastuzumab*: 6 mg/kg dose given intravenously on day 8 of each cycle for patients with HER2-positive breast cancer only
  *8mg/kg loading dose in cycle 1
  HER-2: human epidermal growth factor receptor 2
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
months | 5.6 [4.7 to 6.5]

3. Secondary Outcome: CNS Best Response
Description: CNS best response was defined based on standard criteria. Adding to CR and PR (defined in the primary outcome measure):
  CNS stable disease (SD) is achieving all the following:
  * < 50% reduction in the volumetric sum of all measurable (>/= 1 cm in LD) brain metastases compared to baseline
  * No progression on non-measurable lesions
  * No new CNS lesions (defined as any new lesion >/= 6 mm in LD)
  * Stable or decreasing steroid dose
  * No new/progressive tumor-related neurologic signs or symptoms
  * No progression of extra-CNS disease as assessed by RECIST
  CNS Progressive Disease (PD) was experiencing any of the following:
  ->/- 40% increase in the volumetric sum of all measurable (>/= 1 cm in LD) brain metastases compared to baseline
  * Progression on non-measurable lesions
  * New CNS lesions (defined as any new lesion >/= 6 mm in LD)
  * Increasing steroid dose
  * New/progressive tumor-related neurologic signs or symptoms
  * Progression of extra-CNS disease as assessed by RECIST
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
Participants
  Complete Response | 0
  Partial Response | 24
  Stable Disease >/=24 weeks | 2
  Stable Disease < 24 weeks | 5
  Progressive Disease | 7

4. Secondary Outcome: Site of First Progression
Description: Site of first progression is classified as follows:
  CNS Disease
  * >/=40% increase in the volumetric sum of all measurable lesions as compared to the smallest volume on treatment
  * Progression of non-measurable lesions
  * New lesions (>/=6 mm) Non-CNS Disease
  * Per RECIST 1.0 criteria: PD is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
  Symptomatic
  * Increasing steroid requirement
  * Global deterioration of health status requiring discontinuation of treatment
  * New/progression tumor-related neurologic signs and symptoms (NSS) except for transient worsening lasting </=14 days
Time Frame: Disease was evaluated radiologically at baseline, cycle 2, cycle 4 and thereafter on treatment every 2 cycles (CNS disease) and every 4 cycles (non-disease). Maximum progression follow-up for this study cohort was 18.6 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
participants
  CNS | 15
  Non-CNS | 12
  Both CNS and Non-CNS | 6
  Symptomatic | 2
  No Site | 3

5. Secondary Outcome: Overall Survival
Description: Participants were assessed every 6 months post-treatment. Overall survival is defined as the time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: Maximum survival follow-up for the study cohort was 66 months.
Population: The analysis dataset is comprised of enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
Number analyzed (Participants) | 38
months | 14 [11.7 to 20.7]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed day 1 of each cycle throughout the treatment period. Median (range) treatment duration for this study cohort was 8 cycles (1-20) which approximates months given the 4-week cycle duration.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per NCI Common Toxicity Criteria for Adverse Events version 3 (CTCAEv3). All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | Carboplatin, Bevacizumab, Trastuzumab (if HER2+)
All-Cause Mortality (participants affected / at risk) | 38/38
Serious Adverse Events (participants affected / at risk) | 16/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Bevacizumab, Trastuzumab (if HER2+) (N=38)
Hemoglobin (Blood and lymphatic system disorders) | 1
Ocular-other (Eye disorders) | 1
Fatigue (General disorders) | 6
Leukocytes (Investigations) | 1
Neutrophils (Investigations) | 3
Platelets (Investigations) | 4
ALT, SGPT (Investigations) | 1
AST, SGOT (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Bevacizumab, Trastuzumab (if HER2+) (N=38)
Abdomen, hemorrhage NOS (Gastrointestinal disorders) | 2
Abdomen, pain (Gastrointestinal disorders) | 3
Alkaline phosphatase (Investigations) | 13
Allergic reaction (Immune system disorders) | 3
Allergic reaction (Immune system disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5
ALT, SGPT (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 8
Anxiety (Psychiatric disorders) | 2
AST, SGOT (Investigations) | 23
Ataxia (Nervous system disorders) | 3
Back, pain (Musculoskeletal and connective tissue disorders) | 6
Bone, pain (Musculoskeletal and connective tissue disorders) | 6
Brachial plexopathy (Nervous system disorders) | 1
Breast, pain (Reproductive system and breast disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Buttock, pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Chest/thoracic pain NOS (General disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 2
CNS, hemorrhage (Nervous system disorders) | 2
CNS, hemorrhage (Nervous system disorders) | 4
Cognitive disturbance (Nervous system disorders) | 1
Colon, hemorrhage (Gastrointestinal disorders) | 3
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 14
Constitutional, other (General disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Creatinine (Investigations) | 2
Creatinine (Investigations) | 4
Cushingnoid appearance (Endocrine disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 7
Double vision (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema head and neck (General disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 7
Extremity-lower (gait/walking) (General disorders) | 1
Fatigue (General disorders) | 4
Fatigue (General disorders) | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever w/o neutropenia (General disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Flushing (Vascular disorders) | 1
GI-other (Gastrointestinal disorders) | 4
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 3
Head/headache (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 20
Hemoglobin (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 29
Hot flashes (Vascular disorders) | 2
Hydrocephalus (Nervous system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypercholesterolemia (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 6
Incontinence urinary (Renal and urinary disorders) | 1
Infection Gr0-2 neut, dental-tooth (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 3
Infection Gr0-2 neut, upper airway (Infections and infestations) | 4
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Infection w/ unk ANC sinus (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
INR (Investigations) | 1
Insomnia (Psychiatric disorders) | 2
Jejunum, hemorrhage (Gastrointestinal disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 6
Laryngeal nerve dysfunction (Nervous system disorders) | 1
Larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 5
Leukocytes (Investigations) | 20
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Lymphopenia (Investigations) | 2
Memory impairment (Nervous system disorders) | 2
Mental status (Nervous system disorders) | 2
Metabolic/Laboratory-other (Investigations) | 4
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 2
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Neurologic-other (Nervous system disorders) | 1
Neuropathy CN II vision (Eye disorders) | 1
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 14
Neutrophils (Investigations) | 4
Neutrophils (Investigations) | 20
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic right-side muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 12
Ocular-other (Eye disorders) | 2
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1
Pain-other (General disorders) | 5
Palpitations (Cardiac disorders) | 1
Peripheral arterial ischemia (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1
Platelets (Investigations) | 3
Platelets (Investigations) | 27
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 8
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
PTT (Investigations) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 6
Rigors/chills (General disorders) | 1
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Sinus, pain (Nervous system disorders) | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 4
Speech impairment (Nervous system disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Taste disturbance (Nervous system disorders) | 2
Tearing (Eye disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Tremor (Nervous system disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 2
Visceral arterial ischemia (Vascular disorders) | 3
Vision-blurred (Eye disorders) | 2
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No